CLINICAL TRIAL: NCT00162110
Title: A Phase II Trial of Erbitux for Recurrent and Metastatic Mucinous Gastrointestinal Adenocarcinoma Involving the Peritoneal Surfaces
Brief Title: A Trial of Erbitux for Recurrent and Metastatic Mucinous Gastrointestinal Adenocarcinoma Involving the Peritoneal Surfaces
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-063
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Mucinous Gastrointestinal Adenocarcinoma
MeSH Terms: interventions — Cetuximab

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — mg, IV, 225 mg/m2, weekly, 4-52 weeks depending on response.
  Other Names: Erbitux

SUMMARY:
This is a Phase II open-label trial evaluating the efficacy, and safety of Erbitux in patients with mucinous gastrointestinal adenocarcinoma involving the peritoneal surface.

ELIGIBILITY:
Inclusion Criteria:

* Able to take care of self. Out of bed less than 50% of the day
* Absolute neutrophil count >=1,500
* Platelet count >=100,000
* Total bilirubin count <=1.5 times the upper limit of normal

Exclusion Criteria:

* Prior epidermal growth factor receptor antibody
* Prior treatment with Erbitux
* Other cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of Erbitux in the treatment of mucinous gastrointestinal adenocarcinoma involving the peritoneal surfaces based on clinical response rate.

SECONDARY OUTCOMES:
To evaulate surgically resected tumor specimens of the EGF receptor, mucins 1-6, and anglogenic indices such as vessel counts, VEGF expression, and Ki-67 expression. To evaluate the safety of Erbitux monotherapy in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Local Institution, New York, New York
  - Local Institution, Cincinnati, Ohio